CLINICAL TRIAL: NCT00620776
Title: Combined Treatment for Generalized Anxiety Disorder (GAD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Paul Crits-Christoph, Professor of Psychology in Psychiatry, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 802307; 5R34MH072678-02 (NIH)
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Results first posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2016-12

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Cognitive Behavioral Therapy; Psychotherapy plus medication; Combined treatment
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combined Treatment (Experimental): Patients who receive combined cognitive behavioral therapy (CBT) plus medication (venlafaxine XR, flexibly dosed between 75-225 mg/day) treatment for GAD. CBT was once/week sessions for 12 weeks. Medication continued for the full 6 months.
  Interventions: Behavioral: Cognitive Behavioral Therapy; Drug: Venlafaxine XR
- Venlafaxine XR 75-225 mg alone (Active Comparator): These patients receive only medication treatment for GAD. Patients take venlafaxine (flexibly dosed from 75-225 mg/day) as part of NCT00183274 and are assessed over a 6 month period. Medication continued for the full 6 months.
  Interventions: Drug: Venlafaxine XR

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — This cognitive behavioral therapy for GAD has a cognitive restructuring component and an applied relaxation component. Patients will be educated about the nature of anxiety and be trained in the recognition and monitoring of situational, physiological, cognitive, and behavioral cues associated with anxious responding. They will be guided through copings skill rehearsals in addition to imaginal and in vivo exposure to anxiety cues. This cognitive behavioral treatment will consist of 1 to 1.5 hour sessions of psychotherapy, which will be held once weekly over a period of 12 weeks.
  Arms: Combined Treatment
Drug: Venlafaxine XR — Venlafaxine XR, 75-225 mg/d, oral administration. 14 days at 75 mg/d, 150 mg/d for the remaining 6 months, 225 mg/3 for patients unimproved at week 6, tapered at 75 mg/week (this intervention is provided by protocol 709012).
  Other Names: Effexor extended release

SUMMARY:
The purpose of this study is to conduct a preliminary evaluation of the efficacy of combined medication and psychotherapy for generalized anxiety disorder (GAD). The general goals of the current study are to conduct a late stage treatment development study. The goal of this stage of research is to provide a preliminary answer to the question and to gather data to estimate intervention parameters (e.g., effect size, attrition rates, response rates) that would assist in planning further research.

DETAILED DESCRIPTION:
The specific aims of this study are to collect preliminary data relevant to the following hypotheses:

1. Primary Hypothesis: Acute phase improvement for combined cognitive behavioral therapy (CBT) plus medication will be superior to medication alone.
2. Secondary Hypotheses: Combined CBT plus medication will be superior to medication alone on a number of secondary outcome measures, including the core feature of GAD (worry), depressive symptoms, functional impairment, and quality of life.
3. Additional Exploratory Aim: We will explore the comparative relapse rates for the combined CBT plus medication treatment and the medication alone treatment condition at 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* GAD diagnosis by structured interview
* Hamilton Anxiety Scale score of 18 or less
* Clinical Global Impressions Scale score of at least 4
* Hamilton Depression Scale score of 18 or less
* Hamilton Depression Scale suicide item score less than 2
* Use of an effective form of contraception throughout the s

Exclusion Criteria:

* Hypersensitivity to venlafaxine XR
* History of seizures
* Episode of major depressive disorder in the previous 6 months
* History of any psychotic illness, bipolar disorder, or dementia
* Substance abuse and dependence during the past 6 months
* Other anxiety disorders with the exception of social phobia as long as GAD is primary
* Regular use of anxiolytics or antidepressants within 7 days of study onset
* Use of fluoxetine or monoamine oxidase inhibitors within 28 days of study onset (low dose usage of benzodiazepines will not prevent participation)
* Use of other psychotic medication besides benzodiazepines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2006-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Crits-Christoph, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, 3535 Market Street, Suite 650, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three hundred thirty four patients enrolled in the first phase (6-month open-label) of a parent medication trial for GAD (NCT00183274) were recruited and seen in one of four primary care practices or a psychopharmacology clinic in a university setting from 2005 to 2009. The current study was conducted from October, 2006 to March, 2008.
Pre-assignment Details: Of 334 patients who consented to the parent trial, 66 did not receive study drug (64 withdrew consent and 2 were protocol violators), leaving 268 who received at least one dose of open-label venlafaxine XR. For this study, 77 patients were randomly assigned to be offered CBT and 40 patients to not be offered CBT.
Groups:
- Combined Treatment: Patients received Venlafaxine XR (75-225 mg/d) plus 12 weeks of CBT (one 1 to 1.5 hour session per week) for GAD over a period of 6 months.
- Medication Alone: Patients received Venlafaxine XR (75-225 mg/d) alone as treatment for GAD over a period of 6 months.
Period: Overall Study
Arm/Group | Combined Treatment | Medication Alone
Started | 29 (29 patients (of the 77 that were randomly assigned to add on CBT) consented to this option.) | 40 (All 40 patients that were randomly assigned to not be offered CBT consented to this option.)
Received at Least One Session/Dose | 26 (26 out of 29 that consented to the combined treatment option received at least one session of CBT.) | 35 (35 out of 40 that consented to receive medication alone received at least one dose of medication.)
Completed | 17 (17 out of 26 attended the week 24 (last) assessment.) | 24 (24 out of 35 attended the week 24 (last) assessment.)
Not Completed | 12 | 16
Not completed — Did not receive treatment | 3 | 5
Not completed — Adverse Event | 2 | 3
Not completed — Lack of Efficacy | 2 | 1
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: 26 out of 29 patients who consented to receive combined treatment received at least one session of CBT. 35 out of 40 patients who consented to received medication only received at least one dose of medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined Treatment | Medication Alone | Total
Number analyzed (Participants) | 26 | 35 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (16.0) | 46.6 (19.8) | 47.0 (18.3)
Gender [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 9 | 17 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 24 | 35 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 10 | 18
  White | 17 | 25 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 35 | 61

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Anxiety Rating Scale (HAM-A)
Description: The HAM-A was used to measure the severity of anxiety symptoms. The scale consists of 14 items; each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate and 25-30 moderate to severe anxiety. This measure was conducted by research psychiatrists trained and highly experienced in the use of these scales. The evaluators were blind to group assignment.
Time Frame: Data collected as part of protocol 709012 at baseline, week 2, 4, 6, 8, 12, 16, 20, and 24
Population: Number analyzed at various time points differ due to patient dropout.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Treatment | Medication Alone
Number analyzed (Participants) | 26 | 35
units on a scale
  Baseline | 25.9 (2.6) | 23.8 (2.7)
  Week 2 | 20.9 (5.0) | 19.4 (5.1)
  Week 4: number analyzed (Participants) | 26 | 31
  Week 4 | 17.3 (5.6) | 14.7 (5.6)
  Week 6: number analyzed (Participants) | 26 | 28
  Week 6 | 13.5 (6.5) | 10.9 (5.5)
  Week 8: number analyzed (Participants) | 26 | 27
  Week 8 | 12.7 (7.5) | 7.8 (6.0)
  Week 12: number analyzed (Participants) | 25 | 26
  Week 12 | 10.8 (7.2) | 5.9 (4.3)
  Week 16: number analyzed (Participants) | 20 | 27
  Week 16 | 8.1 (6.9) | 4.3 (3.1)
  Week 20: number analyzed (Participants) | 18 | 25
  Week 20 | 6.2 (5.5) | 4.3 (3.2)
  Week 24: number analyzed (Participants) | 17 | 24
  Week 24 | 6.5 (5.4) | 3.4 (1.9)
Statistical Analysis 1: Comparison: Combined Treatment vs Medication Alone; Mixed model analysis (differential slopes over time) comparing the 26 patients who received combined treatment with at least one CBT session to the 35 patients randomized to venlafaxine XR alone (and received at least one dose) on HAM-A total scores. Only available scores were used (no imputation for missing data). Because the HAM-A demonstrated a relatively rapid improvement early in treatment and then a leveling off, a shifted log-transformation of time of assessment was implemented; Test type: Superiority or Other; p = .17, Mixed Models Analysis

2. Secondary Outcome: Hospital Anxiety Depression Scale (HAD)-Anxiety Score
Description: The HAD was used to assess patients' report of anxiety and depressive symptoms. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. A higher score indicates greater anxiety.
Time Frame: Data collected as part of protocol 709012 at baseline, week 2, 4, 6, 8, 12, 16, 20, and 24
Population: Numbers analyzed at various time points differ due to patient dropout.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Treatment | Medication Alone
Number analyzed (Participants) | 26 | 35
units on a scale
  Baseline | 13.6 (3.4) | 13.0 (4.2)
  Week 2 | 11.7 (4.8) | 10.9 (5.1)
  Week 4: number analyzed (Participants) | 26 | 31
  Week 4 | 10.9 (4.5) | 8.3 (5.0)
  Week 6: number analyzed (Participants) | 26 | 28
  Week 6 | 9.2 (4.7) | 7.1 (4.6)
  Week 8: number analyzed (Participants) | 25 | 27
  Week 8 | 9.0 (4.7) | 5.7 (4.1)
  Week 12: number analyzed (Participants) | 25 | 26
  Week 12 | 6.9 (4.3) | 4.1 (3.4)
  Week 16: number analyzed (Participants) | 20 | 27
  Week 16 | 6.9 (5.2) | 4.6 (3.4)
  Week 20: number analyzed (Participants) | 18 | 24
  Week 20 | 6.2 (4.6) | 4.9 (3.6)
  Week 24: number analyzed (Participants) | 15 | 24
  Week 24 | 6.2 (3.3) | 4.7 (4.5)
Statistical Analysis 1: Comparison: Combined Treatment vs Medication Alone; Analyses were conducted using mixed effects models that tested for differential slopes over time between the CBT plus venlafaxine XR and venlafaxine XR alone groups using only available scores (no imputation for missing data); Test type: Superiority or Other; p = .54, Mixed Models Analysis

3. Secondary Outcome: Hospital Anxiety Depression Scale (HAD)-Depression Score
Description: The HAD was used to assess patients' report of anxiety and depressive symptoms. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. A higher score indicates greater depression.
Time Frame: Data collected as part of protocol 709012 at baseline, week 2, 4, 6, 8, 12, 16, 20, and 24
Population: Numbers analyzed at various time points differ due to patient dropout.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Treatment | Medication Alone
Number analyzed (Participants) | 26 | 35
units on a scale
  Baseline | 9.8 (5.7) | 7.3 (3.4)
  Week 2 | 8.5 (5.1) | 6.8 (3.9)
  Week 4: number analyzed (Participants) | 26 | 31
  Week 4 | 7.9 (5.1) | 5.3 (3.8)
  Week 6: number analyzed (Participants) | 26 | 28
  Week 6 | 6.3 (5.0) | 4.5 (3.3)
  Week 8: number analyzed (Participants) | 25 | 27
  Week 8 | 7.0 (5.3) | 3.4 (3.3)
  Week 12: number analyzed (Participants) | 25 | 26
  Week 12 | 5.5 (4.6) | 2.9 (2.7)
  Week 16: number analyzed (Participants) | 20 | 27
  Week 16 | 5.6 (4.9) | 2.0 (2.3)
  Week 20: number analyzed (Participants) | 18 | 24
  Week 20 | 4.3 (4.3) | 2.1 (2.3)
  Week 24: number analyzed (Participants) | 15 | 24
  Week 24 | 4.7 (3.9) | 2.9 (3.1)
Statistical Analysis 1: Comparison: Combined Treatment vs Medication Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .86, Mixed Models Analysis

4. Secondary Outcome: Hamilton Rating Scale for Depression (HAM-D)-17-item Score
Description: The 17-item version of the HAM-D was used to assess severity of depressive symptoms. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2.The total score is the sum of the 17 items, with a range from 0 to 50. A higher scores indicates greater depression. The ratings were conducted by research psychiatrists trained and highly experienced in the use of these scales. The evaluators were blind to group assignment.
Time Frame: Data collected as part of protocol 709012 at baseline, week 12, and week 24
Population: Numbers analyzed at various time points differ due to patient dropout.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Treatment | Medication Alone
Number analyzed (Participants) | 26 | 35
units on a scale
  Baseline | 13.1 (2.2) | 12.3 (2.8)
  Week 12: number analyzed (Participants) | 23 | 26
  Week 12 | 7.0 (3.4) | 3.9 (2.6)
  Week 24: number analyzed (Participants) | 17 | 24
  Week 24 | 5.1 (4.0) | 3.0 (1.7)
Statistical Analysis 1: Comparison: Combined Treatment vs Medication Alone; Data collected at week 24 were analyzed using analysis of covariance (ANCOVA) with the baseline score as the covariate; Test type: Superiority or Other; p = .051, ANCOVA

5. Secondary Outcome: Clinical Global Impression (CGI)-Severity Score
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale (1=normal; 7 = extremely ill) that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. The ratings were conducted by research psychiatrists trained and highly experienced in the use of these scales. Evaluators were blind to group assignment.
Time Frame: Data collected as part of protocol 709012 at baseline, week 2, 4, 6, 8, 12, 16, 20, and 24
Population: Number analyzed at each time point differs due to patient dropout.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Treatment | Medication Alone
Number analyzed (Participants) | 26 | 35
units on a scale
  Baseline: number analyzed (Participants) | 26 | 34
  Baseline | 4.7 (0.6) | 4.7 (0.5)
  Week 2 | 4.1 (0.6) | 3.9 (0.7)
  Week 4: number analyzed (Participants) | 25 | 31
  Week 4 | 3.6 (0.8) | 3.2 (1.0)
  Week 6: number analyzed (Participants) | 26 | 28
  Week 6 | 3.0 (1.0) | 2.6 (1.0)
  Week 8: number analyzed (Participants) | 26 | 25
  Week 8 | 2.9 (1.3) | 1.9 (1.0)
  Week 12: number analyzed (Participants) | 25 | 26
  Week 12 | 2.4 (1.1) | 1.6 (0.7)
  Week 16: number analyzed (Participants) | 19 | 27
  Week 16 | 2.1 (1.1) | 1.4 (0.6)
  Week 20: number analyzed (Participants) | 17 | 25
  Week 20 | 1.7 (0.9) | 1.4 (0.6)
  Week 24: number analyzed (Participants) | 17 | 24
  Week 24 | 1.8 (1.1) | 1.2 (0.4)
Statistical Analysis 1: Comparison: Combined Treatment vs Medication Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .06, ANCOVA

6. Secondary Outcome: Clinical Global Impression (CGI)-Improvement Score
Description: The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale (1= very much improved; 7 = very much worse) that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. The ratings were conducted by research psychiatrists trained and highly experienced in the use of these scales. Evaluators were blind to group assignment.
Time Frame: Data collected as part of protocol 709012 at baseline, week 2, 4, 6, 8, 12, 16, 20, and 24
Population: Number analyzed at different time points varies due to patient dropout.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Treatment | Medication Alone
Number analyzed (Participants) | 26 | 35
units on a scale
  Baseline: number analyzed (Participants) | 26 | 34
  Baseline | 2.6 (1.9) | 3.1 (1.7)
  Week 2 | 3.3 (0.7) | 3.2 (1.0)
  Week 4: number analyzed (Participants) | 25 | 31
  Week 4 | 2.7 (0.9) | 2.4 (0.8)
  Week 6: number analyzed (Participants) | 26 | 28
  Week 6 | 2.4 (0.9) | 2.0 (0.8)
  Week 8: number analyzed (Participants) | 26 | 25
  Week 8 | 2.3 (1.2) | 1.5 (0.8)
  Week 12: number analyzed (Participants) | 25 | 26
  Week 12 | 1.9 (1.0) | 1.4 (0.6)
  Week 16: number analyzed (Participants) | 19 | 27
  Week 16 | 1.6 (0.8) | 1.2 (0.4)
  Week 20: number analyzed (Participants) | 17 | 25
  Week 20 | 1.4 (0.7) | 1.2 (0.4)
  Week 24: number analyzed (Participants) | 17 | 24
  Week 24 | 1.4 (0.6) | 1.1 (0.3)
Statistical Analysis 1: Comparison: Combined Treatment vs Medication Alone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .95, Mixed Models Analysis

7. Secondary Outcome: Quality of Life Subscale of the General Health Questionnaire (GHQ)
Description: The General Health Questionnaire (GHQ) is a psychometric screening tool to identify common psychiatric conditions. Patients completed the 12 quality of life questions (each on a 0 to 3 scale) on this questionnaire. Scores on the 12 items were added up to create summary score (range = 0 to 36). Higher scores indicate worse health.
Time Frame: Data collected as part of protocol 709012 at baseline, week 12, and week 24
Population: Number analyzed at different time points varies due to patient dropout.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Treatment | Medication Alone
Number analyzed (Participants) | 26 | 35
units on a scale
  Baseline: number analyzed (Participants) | 26 | 33
  Baseline | 34.5 (7.0) | 32.2 (6.4)
  Week 12: number analyzed (Participants) | 25 | 26
  Week 12 | 24.8 (7.3) | 20.4 (5.2)
  Week 24: number analyzed (Participants) | 16 | 23
  Week 24 | 23.8 (6.6) | 22.9 (5.6)
Statistical Analysis 1: Comparison: Combined Treatment vs Medication Alone; Data collected at week 24 were analyzed using ANCOVA with the baseline score as the covariate; Test type: Superiority or Other; p = .17, ANCOVA

8. Secondary Outcome: Penn State Worry Questionnaire (PSWQ)
Description: The Penn State Worry Questionaire is a 16-item inventory that aims to measure the trait of worry, using Likert rating from 1 (not at all typical of me) to 5 (very typical of me). A total score is calculated (range = 16 to 80), with higher scores indicating greater worry.
Time Frame: Data collected as part of protocol 709012 at baseline, week 12, and week 24
Population: Number analyzed at different time points varies due to patient dropout.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Treatment | Medication Alone
Number analyzed (Participants) | 26 | 35
units on a scale
  Baseline: number analyzed (Participants) | 26 | 33
  Baseline | 61.8 (9.5) | 57.9 (12.7)
  Week 12: number analyzed (Participants) | 25 | 26
  Week 12 | 48.6 (11.8) | 42.3 (13.0)
  Week 24: number analyzed (Participants) | 17 | 24
  Week 24 | 46.4 (11.1) | 45.1 (14.0)
Statistical Analysis 1: Comparison: Combined Treatment vs Medication Alone; Data collected at week 24 were analyzed using ANCOVA with the baseline score as the covariate; Test type: Superiority or Other; p = .53, ANCOVA

9. Secondary Outcome: Physical Component Score of the 12-Item Short Form Survey (SF-12)
Description: The Short Form (12) Health Survey is a 12-item, patient-reported survey of patient health. Physical and Mental Health Component Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Data collected as part of protocol 709012 at baseline, week 12, and week 24
Population: Number analyzed at different time points varies due to patient dropout.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Treatment | Medication Alone
Number analyzed (Participants) | 26 | 35
units on a scale
  Baseline: number analyzed (Participants) | 25 | 32
  Baseline | 46.1 (13.6) | 52.7 (10.7)
  Week 12: number analyzed (Participants) | 24 | 26
  Week 12 | 46.2 (12.5) | 51.9 (6.9)
  Week 24: number analyzed (Participants) | 17 | 25
  Week 24 | 45.5 (12.7) | 49.7 (7.0)
Statistical Analysis 1: Comparison: Combined Treatment vs Medication Alone; Data collected at week 24 were analyzed with ANCOVA with baseline data as covariate; Test type: Superiority or Other; p = .23, ANCOVA

10. Secondary Outcome: Mental Component Score of the 12-item Short Form Survey (SF-12)
Description: as for outcome 9
Time Frame: Data collected as part of protocol 709012 at baseline, week 12, and week 24
Population: Number analyzed at different time points varies due to patient dropout.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Combined Treatment | Medication Alone
Number analyzed (Participants) | 26 | 35
units on a scale
  Baseline: number analyzed (Participants) | 25 | 32
  Baseline | 28.5 (9.8) | 31.4 (10.9)
  Week 12: number analyzed (Participants) | 24 | 26
  Week 12 | 46.2 (12.6) | 48.3 (9.5)
  Week 24: number analyzed (Participants) | 17 | 25
  Week 24 | 45.5 (12.7) | 49.8 (10.4)
Statistical Analysis 1: Comparison: Combined Treatment vs Medication Alone; Data collected at week 24 were analyzed with ANCOVA including baseline data as covariate; Test type: Superiority or Other; p = .07, ANCOVA

11. Secondary Outcome: Clinical Response Rate
Description: Clinical response on the HAM-A was defined as a 50% or greater reduction from baseline to last value with the 24-week open label medication phase.
Time Frame: Data collected as part of protocol 709012 at baseline, week 2, 4, 6, 8, 12, 16, 20, and 24
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Treatment | Medication Alone
Number analyzed (Participants) | 26 | 35
Participants | 17 | 25
Statistical Analysis 1: Comparison: Combined Treatment vs Medication Alone; Test type: Superiority or Other; p = .63, Chi-squared

12. Secondary Outcome: 50 Percent or Greater Reduction in PSWQ Score
Description: Clinically significant change was defined on the PSWQ as an estimated (based on linear mixed effects model) endpoint score of less than 50.9. This score was calculated using the PSWQ normative data provided by Gillis, Haaga, and Ford (1995) and the baseline PSWQ mean and standard deviation (SD) from the current sample. The PSWQ mean and SD from the normative and current GAD samples were entered into the Jacobson et al. (1984) formula "c" for clinically significant change. This method provides a cutoff indicating whether or not the level of functioning by a patient is statistically more likely to be in the functional rather than the dysfunctional population.
Time Frame: Data collected as part of protocol 709012 at baseline, week 12, and week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Treatment | Medication Alone
Number analyzed (Participants) | 26 | 35
Participants | 19 | 28
Statistical Analysis 1: Comparison: Combined Treatment vs Medication Alone; Test type: Superiority or Other; p = .52, Chi-squared

ADVERSE EVENTS:
Time Frame: Over the 6-month study period, adverse events were assessed at each visit (from week 2 up to week 24) using an open-ended approach, which was facilitated by the use of a physician-completed medication problem checklist.
Arm/Group | Combined Treatment | Medication Alone
Serious Adverse Events (participants affected / at risk) | 4/26 | 4/35
Other Adverse Events (participants affected / at risk) | 22/26 | 27/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Treatment (N=26) | Medication Alone (N=35)
Severe Fatigue (General disorders) | 2 | 0
Severe Migraine (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Severe Constipation (Gastrointestinal disorders) | 0 | 1
Severe Impact on Libido (General disorders) | 0 | 1
Severe Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Severe Vision Impairment (Eye disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combined Treatment (N=26) | Medication Alone (N=35)
Lightheadedness (General disorders) | 6 | 9
Nausea (Gastrointestinal disorders) | 7 | 6
Diarrhea (Gastrointestinal disorders) | 3 | 3
Muscle Aches (General disorders) | 5 | 4
Insomnia (Psychiatric disorders) | 10 | 6
Headache (General disorders) | 9 | 8
Faintness (General disorders) | 2 | 3
Fatigue (General disorders) | 2 | 3
Decreased Orgasm (General disorders) | 3 | 5
Abdominal Pain (Gastrointestinal disorders) | 2 | 5
Increased Sweating (Endocrine disorders) | 8 | 8
Flatulence (Gastrointestinal disorders) | 5 | 7
Constipation (Gastrointestinal disorders) | 4 | 6
Jittery (General disorders) | 5 | 9
Nightmares/Vivid Dreams (General disorders) | 6 | 4
Anorexia (Psychiatric disorders) | 1 | 2
Anxiety (General disorders) | 0 | 2
Blurred Vision (Eye disorders) | 2 | 1
Decreased Appetite (General disorders) | 2 | 1
Decreased Sex Drive (General disorders) | 5 | 5
Delayed Orgasm (General disorders) | 2 | 1
Drowsiness (General disorders) | 9 | 13
Dry Mouth (General disorders) | 8 | 13
Gas (Gastrointestinal disorders) | 4 | 1
Tremors (General disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
Only one-third of those approached to add on CBT were interested in this option. Strict exclusion criteria reduces the generalizability of the study results. Possible that other forms of CBT treatment may produce different results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No